CLINICAL TRIAL: NCT00467350
Title: Randomized Clinical Trial of Milk and Molasses Enema vs. PEG 3350 for Fecal Impaction in Childhood Constipation
Brief Title: Comparison Trial of Enema vs. PEG 3350 for Constipation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: concern patients in oral cleaout arm had worse outcome
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Melissa Miller, Assistant Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-07-117
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Constipation
Keywords: constipation; treatment; fecal impaction; pediatric
MeSH Terms: conditions — Constipation; Fecal Impaction | interventions — polyethylene glycol 3350; Milk; Enema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enema (Active Comparator): Rectal enema containing mixture of milk and molasses
  Interventions: Drug: milk and molasses enema
- PEG 3350 (Active Comparator): Medication to be taken orally once each day for three consecutive days
  Interventions: Drug: PEG 3350

INTERVENTIONS:
Drug: PEG 3350 — PEG 3350 1.5 gram/kg for disimpaction then 0.8 gram/kg for maintenance
  Other Names: Miralax
  Arms: PEG 3350
Drug: milk and molasses enema — enema 10 cc/kg per rectum (max 500 cc)then PEG 3350 0.8 gram/kg for maintenance
  Other Names: enema
  Arms: enema

SUMMARY:
The purpose of this study is to determine if milk and molasses enema or PEG 3350 works better for treatment of fecal impaction in children who are constipated.

DETAILED DESCRIPTION:
Constipation is a common condition in childhood and occurs without evidence of a pathological condition in most children. Symptoms range from decreased appetite to abdominal pain and constipation is frequently diagnosed in children evaluated in emergency departments. A general guideline for constipation treatment is fecal impaction removal before initiation of maintenance therapy. Disimpaction may be achieved using various oral therapies (e.g. including Polyethylene Glycol 3350 or PEG); however, rectal therapies, most commonly enemas, are frequently used, especially in the emergency/urgent care setting. The optimal treatment has not been established. There are no published randomized studies that compare effectiveness of oral versus rectal treatments.

Comparison: One milk and molasses enema given to the patient in the emergency department compared to three oral doses of PEG 3350 for relief of symptoms due to fecal impaction and constipation.

ELIGIBILITY:
Inclusion Criteria:

* Constipated children who have one of the following three conditions:

  * Fecal impaction (lower quadrant mass or dilated rectum with hard stool),
  * Functional fecal retention (large diameter stools as determined by caregiver <twice/week and retentive behaviors, or
  * Excessive stool in colon on abdominal radiograph as determined by attending radiologist or treating physician

Exclusion Criteria:

* Ill appearing patients (signs of acute surgical abdomen, abnormal vital signs, or overall ill appearing as determined by treating physician)
* Patients whose evaluation in the ED includes more than plain radiographs or urinalysis
* Patients who receive analgesia for the abdominal pain in the ED (except acetaminophen or ibuprofen)
* Non-English speaking patients and families
* Patients with milk allergy
* Patients with molasses allergy
* Patients who are pregnant
* Patients with a chronic medical conditions which may be associated with constipation (including patients with cystic fibrosis, cerebral palsy, hypothyroidism, spinal anomalies, and known gastrointestinal anatomic abnormalities) or a history of prior abdominal or rectal surgery
* Patients who are admitted to an in-patient unit

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K Miller, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample of patients aged 1 to 17 years was recruited between December 2006 and May 2009 from a pediatric emergency department.
Pre-assignment Details: There were no significant events that occurred after enrollment and before study arm assignment.
Period: Overall Study
Arm/Group | Enema | PEG 3350
Started | 41 | 39
Completed | 40 | 39
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enema | PEG 3350 | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (0.7) | 6.9 (0.7) | 6.9 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 14 | 19 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 18 | 30
  African American | 17 | 14 | 31
  Hispanic | 6 | 5 | 11
  other | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Main Symptom Improvement
Description: On day 5, the number of participants who respond "improved" to the question "Has your child's main symptom improved, stayed the same or gotten worse?"
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Enema | PEG 3350
Number analyzed (Participants) | 40 | 39
Participants | 28 | 22
Statistical Analysis 1: Comparison: Enema vs PEG 3350; Test type: Superiority or Other — Similar to previous studies, the main outcome measure was the change in the child's main symptom. Changes were determined by the question "Has your child's main symptom improved, stayed the same or gotten worse?" The main symptom was defined as the chief complaint identified during the triage process. For analysis, responses were dichotomized into 2 groups: improved/better versus worse/same; A χ2 test was used to examine the difference in probabilities of experiencing an outcome between treatment arms and differences were expressed by Mantel-Haenszel common OR estimate with 95% confidence interval (CI)

ADVERSE EVENTS:
Arm/Group | Enema | PEG 3350
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 1/40 | 4/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enema (N=40) | PEG 3350 (N=39)
treatment failure (Gastrointestinal disorders) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
More than half of patients who were approached declined participation. A moderate number of patients (29%) were lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No